CLINICAL TRIAL: NCT01137071
Title: A Phase II Trial of Hu3S193 Consolidation Therapy for Patients With Relapsing Platinum-sensitive Ovarian, Primary Peritoneal and Fallopian Tubes Adenocarcinoma, Who Achieved a Second Complete Response
Brief Title: Consolidation Therapy With Hu3S193 for Women With Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Total number of pts expected to be enrolled would not be met.
Sponsor: Recepta Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCP-Ov-01.10
Record Dates: First submitted 2010-05-31; First posted 2010-06-04 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monoclonal antibody hu3S193 (Experimental): Monoclonal antibody hu3S193 will be administered to 51 patients at the dose of 30mg/m2 every other week (total of 12 infusions) for a total of 23 weeks.
  Interventions: Biological: Monoclonal antibody Hu3S193

INTERVENTIONS:
Biological: Monoclonal antibody Hu3S193 — 30 mg/m2 of Monoclonal antibody Hu3S193, IV as a single agent every two weeks, in a total of 12 doses (treatment period duration: 23 weeks). Anti-Lewis Y humanized monoclonal antibody designated "orphan drug" by the FDA on March 09, 2012 for the treatment of ovarian cancer, not yet approved for the orphan designation.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as Hu3S193, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well Hu3S193 works as a consolidation therapy for women with relapsing platinum-sensitive ovarian, primary peritoneal or fallopian tube cancer.

DETAILED DESCRIPTION:
This is a phase II multicenter trial with Hu3S193 as a single agent in a consolidation strategy in patients with relapsing platinum-sensitive ovarian, primary peritoneal and fallopian tubes cancer who achieve a second Complete Response after a platinum-based chemotherapy after platinum-based chemotherapeutical regimen. Fifty-one (51) patients with relapsing platinum-sensitive ovarian, primary peritoneal or fallopian tubes adenocarcinoma will receive doses of 30 mg/m2 of Hu3S193 as a single agent every two weeks, in a total of 12 doses (treatment period duration: 23 weeks). After the treatment period, patients will be evaluated every 3 months for the first two years, and every 6 months for more 3 years, and then in an annual-basis until disease progression or death, whichever happens first.

ELIGIBILITY:
Inclusion Criteria:

1. The Informed Consent Form (ICF) must be signed before the performance of any study specific procedure or treatment.
2. Female patients of >= 18 years of age.
3. Relapsing ovarian adenocarcinoma, fallopian tubes or primary peritoneal who achieved a complete clinical response after the first treatment of relapse with platinum-based regimen. A complete response is defined as the absence of cancer related symptoms, normal physical exam, normal CA-125 (tumor marker) level, normal chest X-ray and CT-scan of abdomen/pelvis. Eligibility allows the presence of nonspecific findings as long as not showing clear evidence of disease such as: lymph node and/or soft tissue abnormalities <= 1.0 cm which are frequently present on the pelvis and will not be considered to be a conclusive evidence of disease.
4. Expression of antigen Ley documented by immunohistochemistry of archived primary or metastatic tumor samples.
5. The patient must have been submitted at least to hysterectomy and bilateral salpingo-oophorectomy before entering the study and must have received platinum-based chemotherapy as adjunctive or neo-adjunctive treatment at the first presentation.
6. At least 5 and no more than 8 cycles of platinum combination therapy (i.e. doublet) as treatment for the first relapse.
7. All side effects from chemotherapy must have been resolved or must be grade 1.
8. Interval between the last dose of the treatment with platinum that achieved clinical CR (complete response) and the first dose of Hu3S193 =< 8 weeks.
9. Karnofsky performance status >= 70%.
10. Results of laboratorial exams in the first 2 weeks before drug infusion within the following values:

    * Absolute Neutrophil Count >= 1.5 x 10x3 / mm3
    * Platelet count >= 100 x 10x3 / mm3
    * Blood bilirubin <= 2.0 mg/dL
    * Aspartate aminotransaminase (AST) and Alanine aminotransferase (ALT) <= 2.5 x upper limit of normal (ULN).
    * Blood creatinine <= 2.0 mg/dL.
    * Prothrombin time < 1.3 x control
11. Expected survival >= 12 months.
12. Patients must be willing to participate and be able to comply with the protocol throughout the study.

Exclusion Criteria:

1. Mucinous or clear cell histology.
2. Patients must not have received Bevacizumab as part of their treatment on relapse.
3. Diagnosis of primary tumor relapse made exclusively based on elevated levels of serum CA-125 with values <2-fold the upper limit of normality.
4. Concomitant use of systemic corticosteroids or immunosuppressive agents.
5. Known CNS (central nervous system) involvement by tumor.
6. Clinically significant heart disease (New York Heart Association Class III or IV).
7. ECG indicating clinically significant arrhythmia.
8. History of myocardial infarction within 6 months.
9. Other serious diseases, (e.g.: serious infections requiring antibiotics, bleeding disorders, chronic inflammatory bowel disease, or diseases that may interfere in the obtainment of accurate study results).
10. Radiotherapy treatment, radiopharmaceuticals (e.g. 32P), biological therapy, anti-estrogen therapy (including tamoxifen), immunotherapy or surgery within 4 weeks before the first administration of investigational product fail to recover from toxic effects of any of these therapies within 6 weeks prior to study inclusion.
11. Exposure to any investigational product within 4 months prior to study inclusion.
12. Previous treatment with a humanized murine antibody and/or fragment of such antibody.
13. Previous history of tumor (excluding appropriately treated non-melanoma skin cancer or carcinoma in situ of the cervix or no evidence of disease within at least 5 years for previous breast cancer or stage I endometrial cancer).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oren Smaletz, MD, Study Chair — Recepta Biopharma S.A.
Locations (8):
- Brazil (8):
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Cetus Hospital-Dia Oncologia Ltda - Filial Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Fundação Amaral Carvalho, Jaú, São Paulo
  - Instituto do Câncer do Estado de São Paulo "Octávio Frias de Oliveira", São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
Recepta Biopharma understands the importance of individual-patient data (IPD) sharing and will include it in its future clinical studies; however, as this clinical study initiated in Apr-2011, an IPD was not planned.

REFERENCES:
- [Derived] Smaletz O, Ismael G, Del Pilar Estevez-Diz M, Nascimento ILO, de Morais ALG, Cunha-Junior GF, Azevedo SJ, Alves VA, Moro AM, Yeda FP, Dos Santos ML, Majumder I, Hoffman EW. Phase II consolidation trial with anti-Lewis-Y monoclonal antibody (hu3S193) in platinum-sensitive ovarian cancer after a second remission. Int J Gynecol Cancer. 2021 Apr;31(4):562-568. doi: 10.1136/ijgc-2020-002239. Epub 2021 Mar 4. PMID 33664128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Brazilian, multicentric clinical trial. From April 12, 2011 to October 31, 2013 a total of 37 patients were screened for this study, of whom 29 received at least one dose of the investigational product and 07 were considered noneligible.
Pre-assignment Details: Patients were considered included in the study on the day of the first investigational product administration after investigator assured that patients met all the inclusion criterions and none of the exclusion criterions.
Groups:
- hu3S193: hu3S193: 30mg/m2, intravenous, every other week (total of 12 infusions) for a total of 23 weeks
Period: Overall Study
Arm/Group | hu3S193
Started | 29 (all patients considered eligible were included on the study)
Completed | 15 (Of the eligible patients)
Not Completed | 14
Not completed — Disease Progression | 11
Not completed — Withdrawal by Subject | 2
Not completed — Wrongly Included | 1

BASELINE CHARACTERISTICS:
Population: A total of 37 patients were screened for this study of whom 29 were considered eligible and included in the study (baseline participants).
Groups:
- Monoclonal Antibody hu3S193: hu3S193: 30mg/m2, intravenous, every other week (total of 12 infusions) for a total of 23 weeks
Arm/Group | Monoclonal Antibody hu3S193
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: Years] | 55.69 [29 to 67]
Gender [Count of Participants; unit: Participants] — # of Female patients is due to the inclusion criteria number #02: "Female patients of ≥18 years of age"
  Participants
    Female | 29
    Male | 0
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity/Color was recorded at screening
  participants
    White | 24
    Black | 1
    Yellow | 0
    Brown | 4
    Other | 0
Region of Enrollment [Number; unit: participants] — The clinical trial was performed only in Brazil
  participants
    Brazil | 29

OUTCOME MEASURES:

1. Primary Outcome: 1-year PFS2 Rate After the Beginning of Rescue Platinum-based Chemotherapy
Description: PFS2 is defined by the interval from the beginning of rescue platinum-based chemotherapy until documented disease progression or death for any cause while the patient was under study or during the prolonged follow-up period.
  Disease progression is defined by appearance of any new lesion (measurable and non-measurable) by the RECIST criteria. Disease progression date is the date when a new lesion is documented.
Time Frame: 1-Year - From platinum-based rescue chemotherapy start date until documented disease progression or death of any cause whichever occurred first.
Population: In the ITT (intention to treat) population, 25 patients out of the 29 considered for the PFS2 analysis presented disease progression or death and 4 were censored. The median time to disease progression or death was 11.8 months (95% CI (confidence interval), 10.6 to 13.9 months).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Months | 11.7614 [10.5902 to 13.9251]

2. Secondary Outcome: 1-year Disease Progression-free Survival Rate
Time Frame: 1 year from the beginning of platinum-based rescue chemotherapy start date
Population: In the ITT (Intention-to-treat) population, 25 patients out of the 29 considered for the PFS2 analysis presented disease progression or death and 4 were censored.
Measure: Number; unit: percentage of participants
Arm/Group | hu3S193
Number analyzed (Participants) | 29
percentage of participants | 48.2

3. Secondary Outcome: Two-year Overall Survival Rate
Description: Overall survival was calculated as the time interval between the date of beginning of rescue platinum-based chemotherapy and date of death for any cause.
Time Frame: 2-year overall survival rate after the beginning of rescue platinum-based chemotherapy.
Population: Within the ITT population, 7 patients died and 22 were censored. The 2-year overall survival rate was 70.7%.
Measure: Number; unit: percentage of participants
Arm/Group | hu3S193
Number analyzed (Participants) | 29
percentage of participants | 70.7

4. Secondary Outcome: Safety - Vital Signs - Heart Rate
Description: Vital signs were assessed throughout the study treatment (consolidation therapy).Through study completion, an average of 27 weeks.
Time Frame: Baseline, week 2 , week 4 and week 27
Population: All patients enrolled in this study received at least one dose of Hu3S193 (30 mg/m2) - ITT dataset. Baseline n=29, week 2 n=27, week 4 n= 28, week 27 n= 14
Measure: Median (Standard Deviation); unit: bpm
Groups:
- hu3S193: hu3S193 was administered to 29 patients at the dose of 30mg/m2 every other week (total of 12 infusions) for a total of 23 weeks.
Arm/Group | hu3S193
Number analyzed (Participants) | 29
bpm
  Baseline | 78.00 (12.11)
  Week 2 | 80.00 (11.49)
  Week 4 | 76.00 (10.58)
  Week 27 | 75.00 (9.84)

5. Secondary Outcome: Safety - Vital Signs - Respiratory Rate
Description: Vital signs during the study treatment (consolidation therapy). Through study completion, an average of 27 weeks.
Time Frame: Baseline, week 2, week 4 and week 27
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: ipm (Incursions per minute)
Arm/Group | hu3S193
Number analyzed (Participants) | 29
ipm (Incursions per minute)
  Baseline | 19.00 (2.10)
  Week 2 | 19.00 (1.62)
  Week 4 | 19.00 (1.59)
  Week 27 | 19.00 (1.86)

6. Secondary Outcome: Safety - Vital Signs - Systolic and Diastolic Blood Pressure
Description: Both parameters were assessed throughout the study treatment. Vital signs during the study treatment (consolidation therapy). Through study completion, an average of 27 weeks.
Time Frame: Baseline, week 2, week 4 and week 27
Population: All patients enrolled in this study received at least one dose of Hu3S193 (30 mg/m2) - ITT dataset. Diastolic Baseline n=29, week 2 n=27, week 4 n= 28, week 27 n= 14/ Systolic Baseline n=28, week 2 n=27, week 4 n= 28, week 27 n= 14
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | hu3S193
Number analyzed (Participants) | 29
mmHg
  Diastolic Baseline | 80.00 (8.88)
  Diastolic Week 2 | 77.00 (9.04)
  Diastolic Week 4 | 70.00 (7.92)
  Diastolic Week 27 | 80.00 (8.63)
  Systolic Baseline | 115.00 (15.93)
  Systolic Week 2 | 110.00 (14.79)
  Systolic Week 4 | 118.00 (11.32)
  Systolic Week 27 | 120.00 (13.00)

7. Secondary Outcome: Safety - Vital Signs - Temperature
Description: Vital signs during the study treatment (consolidation therapy). Through study completion, an average of 27 weeks.
Time Frame: Baseline, week 2, week 4 and week 27
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: °C
Arm/Group | hu3S193
Number analyzed (Participants) | 29
°C
  Baseline | 36.00 (0.41)
  Week 2 | 36.00 (0.50)
  Week 4 | 35.90 (0.43)
  Week 27 | 35.70 (0.51)

8. Secondary Outcome: Incidence of Adverse Events (AEs) - Gastrointestinal Disorders
Description: The Good Clinical Practice Guidelines define an Adverse Event as any untoward medical event that occurs in a patient or study patient receiving a pharmaceutical product, regardless of its causal relationship with the study treatment. Accordingly, an AE was considered as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or aggravated) temporally associated with the use of an investigational product.
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Nausea | 19
  Vomiting | 17
  Abdominal pain | 9
  Constipation | 7
  Diarrhoea | 6
  Abdominal pain upper | 3
  Dry Mouth | 2
  Dyspepsia | 2
  Abdominal pain lower | 1
  Intestinal Obstruction | 1

9. Secondary Outcome: Incidence of Adverse Events (AEs) - General Disorders and Administration Site Conditions
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Influenza like illness | 8
  Fatigue | 3
  Pain | 2
  Pyrexia | 1

10. Secondary Outcome: Incidence of Adverse Events (AEs) - Musculoskeletal and Connective Tissue Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Myalgia | 4
  Back pain | 3
  Pain in extremity | 2
  Arthralgia | 1
  Groin pain | 1
  Knee pain | 1
  Muscle tightness | 1
  Musculoskeletal pain | 10

11. Secondary Outcome: Incidence of Adverse Events (AEs) - Immune System Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Hypersensitivity | 9
  Drug Hypersensitivity | 2

12. Secondary Outcome: Incidence of Adverse Events (AEs) - Nervous System Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Headache | 9
  Paraesthesia | 1
  Peripheral sensory neuropathy | 1
  Tremor | 1

13. Secondary Outcome: Incidence of Adverse Events (AEs) - Investigations
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Neutrophil count decreased | 5
  White blood cell count decreased | 3

14. Secondary Outcome: Incidence of Adverse Events (AEs) - Respiratory, Thoracic and Mediastinal Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Cough | 6
  Productive Cough | 1

15. Secondary Outcome: Incidence of Adverse Events (AEs) - Infections and Infestations; Gastrointestinal Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Oral Herpes | 2
  Clostridium difficile colitis | 1
  Gastroenteritis | 1
  Tooth abscess | 1

16. Secondary Outcome: Incidence of Adverse Events (AEs) - Blood and Lymphatic System Disorders (Anaemia)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 4

17. Secondary Outcome: Incidence of Adverse Events (AEs) - Infections and Infestations; Respiratory, Thoracic and Mediastinal Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Sinusitis | 2
  Respiratory tract infection | 1
  Tonsillitis | 1

18. Secondary Outcome: Incidence of Adverse Events (AEs) - Psychiatric Disorders (Anxiety)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Groups:
- hu3S193: Monoclonal antibody hu3S193 was administered to 29 patients at the dose of 30mg/m2 every other week (total of 12 infusions) for a total of 23 weeks.
  Anti-Lewis Y humanized monoclonal antibody designated "orphan drug" by the FDA on March 09, 2012 for the treatment of ovarian cancer, not yet approved for the orphan designation.
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 4

19. Secondary Outcome: Incidence of Adverse Events (AEs) - Vascular Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Hypertension | 2
  Hyperaemia | 1
  Hypotension | 1

20. Secondary Outcome: Incidence of Adverse Events (AEs) - Cardiac Disorders; General Disorders and Administration Site Conditions; Respiratory, Thoracic and Mediastinal Disorders (Chest Pain)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 3

21. Secondary Outcome: Incidence of Adverse Events (AEs) - General Disorders and Administration Site Conditions; Musculoskeletal and Connective Tissue Disorders (Chills)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 3

22. Secondary Outcome: Incidence of Adverse Events (AEs) - Skin and Subcutaneous Tissue Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Erythema | 2
  Pruritus | 2

23. Secondary Outcome: Incidence of Adverse Events (AEs) - Ear and Labyrinth Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Cerumen impaction | 1
  Ear pain | 1

24. Secondary Outcome: Incidence of Adverse Events (AEs) - Hepatobiliary Disorders; Injury, Poisoning and Procedural Complications (Hepatotoxicity)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

25. Secondary Outcome: Incidence of Adverse Events (AEs) - Immune System Disorders; General Disorders and Administration Site Conditions; Injury, Poisoning and Procedural Complications (Infusion Related Reaction)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

26. Secondary Outcome: Incidence of Adverse Events (AEs) - Immune System Disorders; Respiratory, Thoracic and Mediastinal Disorders
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Bronchospasm | 1
  Rhinitis allergic | 1

27. Secondary Outcome: Incidence of Adverse Events (AEs) - Musculoskeletal and Connective Tissue Disorders; General Disorders and Administration Site Conditions; Nervous System Disorders (Spinal Pain)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

28. Secondary Outcome: Incidence of Adverse Events (AEs) - Musculoskeletal and Connective Tissue Disorders; Injury, Poisoning and Procedural Complications
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Hip fracture | 1
  Upper limb fracture | 1

29. Secondary Outcome: Incidence of Adverse Events (AEs) - Psychiatric Disorders (Depression)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

30. Secondary Outcome: Incidence of Adverse Events (AEs) - Renal and Urinary Disorders (Dysuria)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

31. Secondary Outcome: Incidence of Adverse Events (AEs) - Renal and Urinary Disorders; Infections and Infestations (Urinary Tract Infection)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

32. Secondary Outcome: Incidence of Adverse Events (AEs) - Reproductive System and Breast Disorders (Vulvovaginal Dryness)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

33. Secondary Outcome: Incidence of Adverse Events (AEs) - Respiratory, Thoracic and Mediastinal Disorders; Cardiac Disorders (Dyspnoea)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 2

34. Secondary Outcome: Incidence of Adverse Events (AEs) - Skin and Subcutaneous Tissue Disorders; Injury, Poisoning and Procedural Complications
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence
  Excoriation | 1
  Injection site erythema | 1

35. Secondary Outcome: Incidence of Adverse Events (AEs) - Cardiac Disorders; Vascular Disorders; Nervous System Disorders (Dizziness)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

36. Secondary Outcome: Incidence of Adverse Events (AEs) - Ear and Labyrinth Disorders; Nervous System Disorders (Vertigo)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

37. Secondary Outcome: Incidence of Adverse Events (AEs) - Endocrine Disorders; Metabolism and Nutrition Disorders (Hyperglycaemia)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

38. Secondary Outcome: Incidence of Adverse Events (AEs) - Eye Disorders (Ocular Hyperaemia)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

39. Secondary Outcome: Incidence of Adverse Events (AEs) - Gastrointestinal Disorders; Infections and Infestations; Respiratory, Thoracic and Mediastinal Disorders (Pharyngitis)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

40. Secondary Outcome: Incidence of Adverse Events (AEs) - Gastrointestinal Disorders; Reproductive System and Breast Disorders; Renal and Urinary Disorders (Pelvic Pain)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

41. Secondary Outcome: Incidence of Adverse Events (AEs) - Gastrointestinal Disorders; Vascular Disorders (Anal Haemorrhage)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

42. Secondary Outcome: Incidence of Adverse Events (AEs) - General Disorders and Administration Site Conditions; Injury, Poisoning and Procedural Complications (Hyperthermia)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

43. Secondary Outcome: Incidence of Adverse Events (AEs) - General Disorders and Administration Site Conditions; Injury, Poisoning and Procedural Complications (Catheter Site Inflammation)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

44. Secondary Outcome: Incidence of Adverse Events (AEs) - Immune System Disorders; Blood and Lymphatic System Disorders; Injury, Poisoning and Procedural Complications (Transfusion Reaction)
Description: The incidence of adverse events (percentage of patients with at least one adverse event and serious adverse events (overall and with reasonable relationship)) was assessed for the safety population
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

45. Secondary Outcome: Incidence of Adverse Events (AEs) - Infections and Infestations; Respiratory, Thoracic and Mediastinal Disorders (Bronchitis)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

46. Secondary Outcome: Incidence of Adverse Events (AEs) - Infections and Infestations; Renal and Urinary Disorders (Urinary Tract Infection Bacterial)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

47. Secondary Outcome: Incidence of Adverse Events (AEs) - Investigations (Blood Cholesterol Increased)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

48. Secondary Outcome: Incidence of Adverse Events (AEs) - Musculoskeletal and Connective Tissue Disorders; General Disorders and Administration Site Conditions; Renal and Urinary Disorders (Flank Pain)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

49. Secondary Outcome: Incidence of Adverse Events (AEs) - Nervous System Disorders; Psychiatric Disorders; Respiratory, Thoracic and Mediastinal Disorders (Hoarseness)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

50. Secondary Outcome: Incidence of Adverse Events (AEs) - Psychiatric Disorders; Nervous System Disorders (Insomnia)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

51. Secondary Outcome: Incidence of Adverse Events (AEs) - Skin and Subcutaneous Tissue Disorders; Infections and Infestations (Tinea Pedis)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

52. Secondary Outcome: Incidence of Adverse Events (AEs) - Skin and Subcutaneous Tissue Disorders; Reproductive System and Breast Disorders (Vulvovaginal Pruritus)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

53. Secondary Outcome: Incidence of Adverse Events (AEs) - Vascular Disorders; Gastrointestinal Disorders (Haemorrhoids)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

54. Secondary Outcome: Incidence of Adverse Events (AEs) - Vascular Disorders; Respiratory, Thoracic and Mediastinal Disorders (Epistaxis)
Description: as for outcome 8
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | hu3S193
Number analyzed (Participants) | 29
Incidence | 1

55. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) - Gastrointestinal Disorders
Description: A SAE was defined as an AE that met one of the following conditions: Death during the protocol-defined surveillance period; Potentially fatal event (defined as a patient at immediate risk of death at the time of the event); An event requiring the patient's hospitalization or prolongation of an existing hospitalization during the protocol-defined surveillance period; An event resulting in congenital anomaly or birth defect; An event resulting in a persistent or significant disability/incapacity; Any other major medical event that did not result in death, was not life threatening, or did not require hospitalization, but that could be considered a SAE when, based on the appropriate medical judgment, it presented a risk for the patient and required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | Monoclonal Antibody hu3S193
Number analyzed (Participants) | 29
Incidence
  Intestinal obstruction | 1
  Vomiting | 1

56. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) - Musculoskeletal and Connective Tissue Disorders - Hip Fracture
Description: as for outcome 55
Time Frame: From the first infusion of medication to 30 days after the last one
Population: All patients who received at least one dose of investigational product were included in the safety dataset.
Measure: Number; unit: Incidence
Arm/Group | Monoclonal Antibody hu3S193
Number analyzed (Participants) | 29
Incidence | 1

57. Secondary Outcome: Overall Mean Pharmacokinetic (PK) Data (Minimum and Maximum Concentrations)
Description: Cmax = Peak (postdosing) Hu3S193 plasma concentration. Cmin = Trough (predosing) Hu3S193 plasma concentration (Cmin). Plasma concentration of Hu3S193 expressed in μg/mL.
Time Frame: Predose and Postdose on weeks 1, 2, 3, 4, 5, 7 and 9
Population: PK samples were analyzed from 10 patients. Dose: 30 mg/m2 every two weeks
Measure: Mean (Standard Deviation); unit: (µg/mL)
Groups:
- Pharmacokinetic: All patients enrolled in the study that received at least 9 doses of investigational product were considered to this analysis.
Arm/Group | Pharmacokinetic
Number analyzed (Participants) | 10
(µg/mL)
  Cmin | 2.14 (0.92)
  Cmax | 18.32 (5.66)

58. Secondary Outcome: Two-year Overall Survival: Median Time to Death
Description: as for outcome 3
Time Frame: 2-year overall survival rate after the beginning of rescue platinum-based chemotherapy.
Population: Within the ITT population, 7 patients died and 22 were censored. The median time to death was 25.1 months (95% CI, 16.7 to 32.4 months).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | hu3S193
Number analyzed (Participants) | 29
months | 25.1 [16.7 to 32.4]

ADVERSE EVENTS:
Time Frame: They were collected from first application of treatment to 30 days after last. Ongoing AEs were followed up until resolution, start of a new treatment, at the investigator discretion or if they became chronic.
Description: After the 30-day period, the investigator reported the adverse events that in his/her opinion were related to investigational product. In this study, AEs terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA) at the Preferred Term (PT) and System Organ Class (SOC) levels.
Arm/Group | hu3S193
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hu3S193 (N=29)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hu3S193 (N=29)
Nausea (Gastrointestinal disorders) | 19 (69)
Vomiting (Gastrointestinal disorders) | 17 (64)
Abdominal pain (Gastrointestinal disorders) | 9 (16)
Constipation (Gastrointestinal disorders) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Influenza like illness (General disorders) | 8 (9)
Fatigue (General disorders) | 3 (4)
Pain (General disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5)
Hypersensitivity (Immune system disorders) | 9 (9)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Headache (Nervous system disorders) | 9 (26)
Neutrophil count decreased (Investigations) | 5 (6)
White blood cell count decreased (Investigations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (14)
Oral herpes (Infections and infestations) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Sinusitis (Infections and infestations) | 2 (3)
Anxiety (Psychiatric disorders) | 4 (8)
Hypertension (Vascular disorders) | 2 (2)
Chest pain (Cardiac disorders) | 3 (4)
Chills (General disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Hepatotoxicity (Hepatobiliary disorders) | 2 (3)
Infusion related reaction (Immune system disorders) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (3)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less